CLINICAL TRIAL: NCT05176769
Title: The Usefulness of Artificial Intelligence for Automated Extraction and Processing of Clinical Data From Electronic Medical Records (CardioMining-AI)
Brief Title: Artificial Intelligence for Automated Clinical Data Exploration From Electronic Medical Records (CardioMining-AI)
Status: Recruiting | Type: Observational
Sponsor: AHEPA University Hospital (Other)
Collaborators: Hippokration Hospital Athens (Unknown); General Hospital of Larissa (Other); University Hospital, Alexandroupolis (Other); University General Hospital of Patras (Other); University General Hospital of Heraklion (Other); George Papanicolaou Hospital (Other); Ippokrateio General Hospital of Thessaloniki (Other)
Responsible Party: Principal Investigator, George Giannakoulas, Associate Professor in Cardiology, AHEPA University Hospital
Other Study IDs: 545/19.11.2021
Record Dates: First submitted 2021-11-24; First posted 2022-01-04 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Artificial Intelligence; Machine Learning; Electronic Medical Records
Keywords: artificial intelligence; machine learning; medical records; digital health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to highlight the usefulness of artificial intelligence and machine learning to develop computer algorithms that will achieve with great reliability, speed and accuracy the automatic extraction and processing of large volumes of raw and unstructured clinical data from electronic medical files.

DETAILED DESCRIPTION:
Despite the rapid development of medicine and computer science in recent years, the medical treatment in modern clinical practice is often empirical and based on retrospective data. With the growing number of patients and their concentration in large tertiary centers, it becomes attractive to systematically collect clinical data and apply them to risk stratification models. However, with the increasing volume of data, manual data collection and processing becomes a challenge, as this approach is time consuming and costly for the healthcare systems. In addition, unstructured information, such as clinical notes, are very often written as free text that is unsuitable for direct analysis. The use of artificial intelligence is very promising and is going to rapidly change the future of medicine in the upcoming years. Due to the automated processes it offers, it is possible to quickly and reliably extract data for further processing. The results from its use can be easily extended to different healthcare systems, amplifying the knowledge produced and improving diagnostic and therapeutic accuracy, and ultimately positively affecting health services. Collecting the vast amount of data from different sources without compromising patients' personal data is a major challenge in modern science.

Electronically-registered clinical notes of patients who were hospitalized in the Cardiology ward of tertiary hospitals will be retrospectively collected, as well as additional files such as the laboratory and imaging examinations related to each hospitalization. Given the size of the participating clinics and the years during which the recording of electronic hospital records in electronic form was applied, it is estimated that the sample of patient records will be about 60.000. All information that could potentially be used to identify a person, such as name, ID number, postal code, place of residence, occupation, will be deleted from these electronic files. Only the age will be recorded, not the exact date of birth of each patient. Only the days of hospitalization will be recorded and not the exact dates of admission and discharge from the hospital. Thus, the data will not be able to be assigned to a specific subject, as no additional information or identifiers will be collected for the subjects. After the files are anonymized, each patient's clinical note will be linked with a specific key ("identifier"). The electronic file that contains the correlation of the "identifier" with the patient's clinical note will be stored in a secure hospital electronic location. The fully anonymized files will initially be manually analyzed to extract information into a database containing all of patients' clinical information, such as discharge diagnoses, medications, treatment protocols, laboratory and diagnostic tests. At the same time, a sample (1/3) of the clinical notes will be analyzed to identify the keywords or phrases associated with each diagnosis (for example, the atrial fibrillation diagnosis will probably be recorded as "atrial fibrillation", " AF ", etc.). By using this generated dictionary of keywords and by integrating artificial intelligence methods and text mining, such as natural language processing (NLP), an automated extraction of data and diagnoses from these electronic medical notes will be attempted. The reliability and accuracy of the computational methods will be evaluated internally, comparing the data extracted automatically with those recorded manually. In addition, the reliability and accuracy of these computational methods will be evaluated externally, applying these methods to 2/3 of the clinical notes in which no association between keywords and specific diagnoses was attempted.

Regarding Greece, the present study aims to be the first to analyze the usefulness of artificial intelligence for automated extraction and processing of unstructured clinical data from patients' medical clinical notes. The results of this study will have a positive impact on:

1. the automation of large-scale data analysis and processing procedures
2. the rapid epidemiological recording and utilization of clinical data
3. the early diagnosis of diseases
4. the development of phenotypic patient profiles that could benefit from targeted therapies
5. the development of clinical decision support systems that will provide information about the possible clinical course of patients after hospital discharge and assist medical decisions
6. the development and validation of prognostic models for major cardiovascular diseases

ELIGIBILITY:
Inclusion Criteria:

* Hospitalised patients in Cardiology Departments in Greece
* Patients whose medical records are electronically stored in each hospital's computer/information systems

Exclusion Criteria:

* Patients that died during hospitalization, and thus no discharge letter was issued

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who were hospitalized in the Cardiology ward of tertiary hospitals and have available electronically-stored clinical notes/hospitalization documents will be included in the study .
Sampling Method: Non-Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of artificial intelligence to automatically extract clinical data from patients' medical records compared with traditional manual data extraction methods | 1 year
  Rate of accurate extraction of clinical data (medical history, discharge diagnoses, medication, etc.) from unstructured clinical notes using automated artificial intelligence methods compared with traditional methods of manual data extraction

SECONDARY OUTCOMES:
Time to all-cause mortality | up to 8 years (from hospital discharge until study primary completion date)
  Length of time (months) until death from any cause during the follow-up period
Time to incident major cardiovascular diseases | up to 8 years (from hospital discharge until study primary completion date)
  Length of time (months) until development of heart failure, diabetes mellitus or coronary artery disease during the follow-up period
Time to rehospitalization for cardiovascular reasons | up to 8 years (from hospital discharge until study primary completion date)
  Length of time (months) until rehospitalization for cardiovascular reasons during the follow-up period
Time to stroke or systemic embolism | up to 8 years (from hospital discharge until study primary completion date)
  Length of time (months) until stroke or systemic embolism during the follow-up period
Time to acute coronary syndrome | up to 8 years (from hospital discharge until study primary completion date)
  Length of time (months) until acute coronary syndrome during the follow-up period

CONTACTS AND LOCATIONS:
Locations (9):
- Greece (9):
  - University Cardiology Clinic, Democritus University of Thrace, Alexandroupoli
  - 1st Department of Cardiology, Hippokration General Hospital, Athens
  - Department of Cardiology, Heraklion University Hospital, Heraklion
  - University General Hospital of Larissa, University of Thessaly, Larissa
  - Department of Cardiology, University of Patras Medical School, Pátrai
  - 1st Cardiology Department, AHEPA University Hospital, Thessaloniki
  - 3rd Cardiology Department, Hippokration Hospital, Thessaloniki
  - Cardiology Department, George Papanikolaou General Hospital, Thessaloniki
  - Laboratory of Medical Physics, Aristotle University of Thessaloniki, Thessaloniki

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analysis plan and results will become available through publications. The analytic code will become available in open source communities/repositories
Supporting Information: Study Protocol, SAP, Analytic Code

REFERENCES:
- [Background] Johnson KW, Torres Soto J, Glicksberg BS, Shameer K, Miotto R, Ali M, Ashley E, Dudley JT. Artificial Intelligence in Cardiology. J Am Coll Cardiol. 2018 Jun 12;71(23):2668-2679. doi: 10.1016/j.jacc.2018.03.521. PMID 29880128
- [Background] Krittanawong C, Zhang H, Wang Z, Aydar M, Kitai T. Artificial Intelligence in Precision Cardiovascular Medicine. J Am Coll Cardiol. 2017 May 30;69(21):2657-2664. doi: 10.1016/j.jacc.2017.03.571. PMID 28545640
- [Background] Madani A, Arnaout R, Mofrad M, Arnaout R. Fast and accurate view classification of echocardiograms using deep learning. NPJ Digit Med. 2018;1:6. doi: 10.1038/s41746-017-0013-1. Epub 2018 Mar 21. PMID 30828647
- [Background] Boag W, Doss D, Naumann T, Szolovits P. What's in a Note? Unpacking Predictive Value in Clinical Note Representations. AMIA Jt Summits Transl Sci Proc. 2018 May 18;2017:26-34. eCollection 2018. PMID 29888035
- [Background] Hashir M, Sawhney R. Towards unstructured mortality prediction with free-text clinical notes. J Biomed Inform. 2020 Aug;108:103489. doi: 10.1016/j.jbi.2020.103489. Epub 2020 Jun 25. PMID 32592755
- [Background] Diller GP, Kempny A, Babu-Narayan SV, Henrichs M, Brida M, Uebing A, Lammers AE, Baumgartner H, Li W, Wort SJ, Dimopoulos K, Gatzoulis MA. Machine learning algorithms estimating prognosis and guiding therapy in adult congenital heart disease: data from a single tertiary centre including 10 019 patients. Eur Heart J. 2019 Apr 1;40(13):1069-1077. doi: 10.1093/eurheartj/ehy915. PMID 30689812
- [Derived] Samaras A, Bekiaridou A, Papazoglou AS, Moysidis DV, Tsoumakas G, Bamidis P, Tsigkas G, Lazaros G, Kassimis G, Fragakis N, Vassilikos V, Zarifis I, Tziakas DN, Tsioufis K, Davlouros P, Giannakoulas G; CardioMining Study Group. Artificial intelligence-based mining of electronic health record data to accelerate the digital transformation of the national cardiovascular ecosystem: design protocol of the CardioMining study. BMJ Open. 2023 Apr 3;13(4):e068698. doi: 10.1136/bmjopen-2022-068698. PMID 37012018